CLINICAL TRIAL: NCT01006785
Title: Phase II Clinical Study: A Randomized, Open, and Dose Ranging Study to Evaluate the Efficacy and Safety of DLBS1425 in Subjects With Metastatic / Advanced Breast Cancer
Brief Title: Efficacy and Safety of DLBS1425 in Subjects With Advanced/Metastatic Breast Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: The study was terminated due to difficulty of find eligible subjects
Sponsor: Dexa Medica Group (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DLBS1425-0209
Record Dates: First submitted 2009-11-01; First posted 2009-11-03 (Estimated); Last update posted 2012-10-18 (Estimated); Status verified 2012-10

CONDITIONS: Breast Cancer
Keywords: Breast Cancer; DLBS 1425; Cancer; Advanced/Metastatic (Stage IIIB/IV) Breast Cancer
MeSH Terms: conditions — Breast Neoplasms; Neoplasms; Neoplasm Metastasis | interventions — DLBS 1425

ARMS (2):
- Treatment I (Experimental): DLBS1425 150 mg three times daily
  Interventions: Drug: DLBS1425
- Treatment II (Experimental): DLBS1425 300 mg three times daily
  Interventions: Drug: DLBS1425

INTERVENTIONS:
Drug: DLBS1425 — 3 X 150 mg daily for 12 - 16 weeks of treatment
  Arms: Treatment I
Drug: DLBS1425 — 3 X 300 mg daily for 12 - 16 weeks of treatment
  Arms: Treatment II

SUMMARY:
The purposes of this study are :

* to investigate the safety and clinical efficacy of sole therapy with DLBS1425 in suppressing disease-(tumour) progression in subjects with advanced/metastatic breast cancer; and
* to determine the minimal effective and safe dose of DLBS1425 in the therapy of advanced/metastatic breast cancer

ELIGIBILITY:
Inclusion Criteria:

* Subjects diagnosed with Stage IIIB or IV breast cancer who have failed with or refuse to receive standard chemotherapies
* Subjects with the expression of ER/PR negative; or positive ER/PR expression but have failed with or refuse to receive hormonal therapy
* Either + or - expression of HER-2/neu gene
* ECOG status = 0-2
* At least have 1 evaluable and measurable metastatic lesion as defined by RECIST criteria
* Adequate haematological, liver, and renal function
* At least 3 weeks has elapsed since prior chemotherapy, radiotherapy, biological/hormonal therapy
* At least 4 weeks has elapsed since surgical biopsy / major surgery

Exclusion Criteria:

* Allergic to the trial product
* Any other disease state, including infections or uncontrolled illnesses that could interfere with trial participation or trial evaluation
* Concurrent herbal (alternative) medicine or food supplements suspected to have effect on cancer disease

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2009-08; Primary Completion 2012-03 (Actual); Study Completion 2012-03 (Actual)

PRIMARY OUTCOMES:
Best overall response rate: proportion of subjects with either complete or partial response according to the Response Evaluation Criteria In Solid Tumors (RECIST) criteria at the end of study | 12 -16 weeks

SECONDARY OUTCOMES:
Time point overall response rate | 6 weeks
Routine hematology | at interval of 2 weeks over the 12 -16 weeks of treatment
  Routine hematology including hemoglobin, hematocrit, red blood cells, white blood cells, differentiation of WBC, and platelet count
Liver function | at interval of 2 weeks over the 12 -16 weeks of treatment
  Liver function including alkaline phosphatase, serum ALT, serum AST, and bilirubin
Renal function | at interval of 2 weeks over the 12 -16 weeks of treatment
  Renal function including serum creatinine
ECHO | at baseline and at week 6, 12, and 16 of treatment
Adverse events | during 12 - 16 weeks of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Abdul Muthalib, Prof. Dr., Principal Investigator — Division of Medical Haematology and Oncology, Department of Internal Medicine, Faculty of Medicine, University of Indonesia / Dr. Cipto Mangunkusumo Hospital
Locations (3):
- Indonesia (3):
  - Dr. Sardjito Hospital, Department of Internal Medicine, Yogyakarta, DI Yogyakarta
  - Dr. Cipto Mangunkusumo Hospital, Division of Medical Haematology and Oncology, Jakarta, DKI Jakarta
  - Dr. Hasan Sadikin Hospital, Department of Internal Medicine, Bandung, West Java